CLINICAL TRIAL: NCT01734291
Title: Brief Multifamily Psychoeducation for Families of Patients With Chronic Major Depression: A Randomized Controlled Trial
Brief Title: Brief Multifamily Psychoeducation for Families of Patients With Chronic Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nagoya City University (Other)
Responsible Party: Principal Investigator, Fujika Katsuki, Associate Professor, Nagoya City University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCUPsychiatricNursing001; ID24593499 (Other Grant/Funding Number: Grants-in-Aid for Scientific Research)
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
Keywords: Family psychoeducation; Major depressive disorder; Family burden
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family psychoeducation plus TAU (Active Comparator): Family psychoeducational therapy in addition to treatment as usual for the patients.
  Interventions: Behavioral: Family psychoeducation
- Treatment as usual(TAU) (Placebo Comparator): Treatment as usual administered by physician and counseling administered by nurse.
  Interventions: Behavioral: Family psychoeducation

INTERVENTIONS:
Behavioral: Family psychoeducation — Family psychoeducational therapy every two weeks for six weeks in addition to treatment as usual administered by physicians

SUMMARY:
The purpose of this study is to examine the effectiveness of brief multifamily psychoeducation to relieve the psychological distress of families of patients with chronic major depression and to improve their family functioning.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a long-lasting illness with significant effects on the patient's family, social life, and work life. Treatment failure results in a low recovery rate and frequent relapses.

Relatives of patients with MDD are fraught with heavy psychosocial burden and show increased rates of depression and anxiety. Among relatives of patients with MDD, the patient's behavior and mood disturbance and relative's emotional distress were associated with the relatives' burden.

Family psychoeducation is recognized as part of the optimal treatment for patients with psychotic disorder. This intervention has been shown to reduce the rates of relapse and hospitalization among individuals with psychotic disorders and is recognized as an evidenced-based treatment for psychotic disorder. Several randomized controlled trials have found that family psychoeducation is effective in enhancing the course of bipolar disorder. However, there are few studies on psychoeducation of families of patients with MDD.

The purpose of this study is to examine the effectiveness of brief multifamily psychoeducation to relieve the psychological distress of families of patients with chronic major depression and to improve their family functioning, in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the criteria for Major Depressive Disorder (MDD) according to DSM-IV.
2. Receives antidepressant therapy.
3. The patient had the first episode of MDD more than one year ago.
4. Currently fulfills the diagnostic threshold for major depressive episode or partial remission.
5. The patient and their family member(s) are aged between 18 and 85 years.
6. The patient has lived with his/her family at the time of participating in this study and is expected to live with his/her family during the investigation period.

Exclusion Criteria:

1. Patients who undergo electroconvulsive therapy (ECT) during the investigation period.
2. Patients who are at serious suicidal risk.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2016-06-20 (Actual); Study Completion 2016-10-09 (Actual)

PRIMARY OUTCOMES:
The change of total score of K6 of family members | The base line, 8, 16 and 32
  The K6 questionnaire is a six-item self-report questionnaire that was developed to screen for DSM-IV depressive and anxiety disorder.

SECONDARY OUTCOMES:
The change of total score of Family Attitude Scale(FAS) of family members | The base line, 8, 16 and 32
  The Family Attitude Scale(FAS) is a 30-item self report inventory and measures families' Expressed Emotion(EE).

CONTACTS AND LOCATIONS:
Overall Officials: Fujika Katsuki, Dr, Principal Investigator — Nagoya City University, School of Nursing
Locations (1):
- Fujika Katsuki, Nagoya, Aichi-ken, Japan

REFERENCES:
- [Background] Katsuki F, Takeuchi H, Watanabe N, Shiraishi N, Maeda T, Kubota Y, Suzuki M, Yamada A, Akechi T. Multifamily psychoeducation for improvement of mental health among relatives of patients with major depressive disorder lasting more than one year: study protocol for a randomized controlled trial. Trials. 2014 Aug 12;15:320. doi: 10.1186/1745-6215-15-320. PMID 25118129
- [Derived] Katsuki F, Takeuchi H, Inagaki T, Maeda T, Kubota Y, Shiraishi N, Tabuse H, Kato T, Yamada A, Watanabe N, Akechi T, Furukawa TA. Brief multifamily Psychoeducation for family members of patients with chronic major depression: a randomized controlled trial. BMC Psychiatry. 2018 Jun 22;18(1):207. doi: 10.1186/s12888-018-1788-6. PMID 29929495